CLINICAL TRIAL: NCT05852535
Title: Spontaneous Evisceration of Infantile Umbilical Hernia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ahmed Kamel Ali Mohamed (Other)
Responsible Party: Sponsor-Investigator, Ahmed Kamel Ali Mohamed, Mr., Assiut University
Organization: Assiut University (Other)
Other Study IDs: AKA171292
Record Dates: First submitted 2023-04-24; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Pediatric Disorder
MeSH Terms: interventions — Space Flight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- case report
  Interventions: Procedure: Exploration

INTERVENTIONS:
Procedure: Exploration — abdominal exploration

SUMMARY:
Infantile umbilical hernia is common in children. It has a regressive course in most cases. Conservative management is the standard in most cases before the age of 3 years unless there are complications such as incarceration, rupture with evisceration which are extremely rare and warrants emergency surgery.

We present a rare case of a 6-month-old child with sudden spontaneous evisceration of infantile umbilical hernia.

DETAILED DESCRIPTION:
Infantile umbilical hernia is common in children. It has a regressive course in most cases. Conservative management is the standard in most cases before the age of 3 years unless there are complications such as incarceration, rupture with evisceration which are extremely rare and warrants emergency surgery.

We present a rare case of a 6-month-old child with sudden spontaneous evisceration of infantile umbilical hernia.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric group

Exclusion Criteria:

* Adult group

Ages: 1 Month to 3 Years | Sex: Male
Age Groups: Child
Study Population: pediatric age group
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2023-05-07 (Estimated); Primary Completion 2023-05-23 (Estimated); Study Completion 2023-05-24 (Estimated)

PRIMARY OUTCOMES:
hospital stay | From April 1, 2023 to April 1, 2024
  hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Ali, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes